CLINICAL TRIAL: NCT06795269
Title: EFFECT OF CRYOTHERAPY ON KINEMATIC GAIT PARAMETERS IN PATIENTS WITH CHRONIC PATELLOFEMORAL PAIN SYNDROME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Makarious Adel Anwar, Physiotherapist specialist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/004880
Record Dates: First submitted 2025-01-16; First posted 2025-01-28 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2023-10

CONDITIONS: CHRONIC PATELLOFEMORAL PAIN SYNDROME
Keywords: Cryotherapy; compression cryotherapy; Biodex Gait Trainer
MeSH Terms: interventions — Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A (control group) (Active Comparator): Thirty patients with PFPS, Their ages ranging from 18 to 40 years old ,Their BMI was from 20 to 25 kg/m2 received treatment in form of Traditional treatment (Strengthening exercise, Stretching, ultrasound and electrotherapy). The treatment performed three time a week for 4 weeks
  Interventions: Other: Conservative treatment
- Group B (Study group) (Experimental): Thirty patients with PFPS, Their ages ranging from 18 to 40 years old ,Their BMI was from 20 to 25 kg/m2 received treatment in form of Traditional treatment (Strengthening exercise, Stretching, ultrasound and electrotherapy) with cryotherapy, The treatment performed three time a week for 4 weeks.
  Interventions: Device: Cryotherapy Compression Machine

INTERVENTIONS:
Device: Cryotherapy Compression Machine — The Cryo Pro is a simple to use cold compression therapy product that requires only ice, water and power. It's unique design is convenient to use, provides pain relief and reduces swelling and inflammation, making recovery faster.
  Arms: Group B (Study group)
Other: Conservative treatment — Strength and stretch exercises for hip and knee large groups of muscles.
  Arms: Group A (control group)

SUMMARY:
this study show the EFFECT OF CRYOTHERAPY ON KINEMATIC GAIT PARAMETERS IN PATIENTS WITH CHRONIC PATELLOFEMORAL PAIN SYNDROME and review its reliability.

Participants were randomly allocated into two equal groups (A and B ) were done by a blinded independent researcher who opened enclosed envelopes containing computer generated randomization serially number index cards using statistical package for social science (SPSS),program (version 20 for windows ,spss, Chicago Illinois,USA) There were no dropouts among the participants throught the study after randomization.

DETAILED DESCRIPTION:
Sixty patients from both genders were participated in this study. they were selected from the outpatient clinic of Faculty of Physical Therapy ,Cairo University with a PFPS.

The Patients of both genders with their ages were ranging from 18 to 40 years old and their BMI was from 20 to 25 kg/m2.

Thirty patients with PFPS, Their ages ranging from 18 to 40 years old ,Their BMI was from 20 to 25 kg/m2 received treatment in form of Traditional treatment (Strengthening exercise, Stretching, ultrasound and electrotherapy). The treatment performed three time a week for 4 weeks.

Thirty patients with PFPS, Their ages ranging from 18 to 40 years old ,Their BMI was from 20 to 25 kg/m2 received treatment in form of Traditional treatment (Strengthening exercise, Stretching, ultrasound and electrotherapy) with cryotherapy, The treatment performed three time a week for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* The patients were diagnosed as patellofemoral pain by an orthopedist.
* The participants were eligible to be included if they had bilateral PFPS or unilateral PFPS.
* Duration of knee pain is 4-5 weeks during 6 months prior to study. (Collins et al., 2010).
* Their ages were ranging from 18 to 40 years (Clin Rheumatol et al., 2012).
* Their BMI was ranging from(20 to 25 kg/m2) (Fischer et al., 2009)

Exclusion Criteria:

* • Rheumatoid Arthritis or other systemic rheumatic diseases.

  * Dementia, psychosis.
  * Active substance abuse disorder; acute or chronic disease, injury, deformity.
  * Operation of the lower limb and knee.
  * Severe hearing or visual impairment.
  * Hospitalization for a cardiovascular condition, cerebral infarction or arrhythmia in the previous 3 months.
  * Recent history of 3 or more falls.
  * Current participation in another OA intervention study.
  * Uncontrolled diabetes mellitus.
  * Intra-articular knee injections in the previous 6 months.
  * Contraindications to cryotherapy application those that feel a high level of discomfort or pain during the application.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-08 (Actual); Primary Completion 2024-10-08 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
Biodex Gait Trainer | 4 weeks
  treadmill with real-time step length visualization (where the foot was placed) was used to assess the selected spatiotemporal gait parameters. During the test, the patient was visually informed about the suggested foot placement/planned length of the step. This three-minute extended test was conducted before and after the rehabilitation program.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy College of Cairo University, Giza, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided